CLINICAL TRIAL: NCT05553964
Title: Prospective, Multi-Center, Non-Randomized Study to Evaluate the 3EO Health SARS-CoV-2 Molecular Diagnostic Test
Brief Title: SARS-CoV-2 OTC At Home Test
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Further usability assessment needed.
Sponsor: 3EO Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3EO-CoV2-01
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — In Vitro Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Study Groups (Experimental): Positives: Symptomatic vs. Asymptomatic Negatives: Symptomatic vs. Asymptomatic
  Each broken down by age groups:
  2-14 years old 15-24 years old 25-64 years old 65+ years old
  Interventions: Diagnostic Test: In Vitro

INTERVENTIONS:
Diagnostic Test: In Vitro — In vitro diagnostic test for COVID-19 using anterior nasal swabs.

SUMMARY:
The objective of this study is to evaluate the 3EO Health COVID-19 Test in individuals presenting at a medical facility. In eligible subjects, nasal samples will be collected for use with the 3EO Health COVID-19 Test, which will be compared to the Zymo® rRT-PCR test results obtained via samples specified by the manufacturer (e.g., AN [anterior nares] swab) to determine accuracy of the 3EO Health COVID-19 Test in detecting COVID-19 in participants.

DETAILED DESCRIPTION:
3EO Health, Inc. has developed the 3EO Health COVID-19 Test, a unique rapid molecular test system, to detect SARS-CoV-2 virus in the OTC setting using a dedicated test reader "3EO Cube" to test nasal swab samples. Early testing will help to determine limit of detection (LOD) of the 3EO Health COVID-19 Test and will be compared to a sensitive molecular test that has been authorized for emergency use by the FDA. The 3EO Health COVID-19 Test will leverage the processing and testing of the 3EO Health Swab device when inserted directly into the reaction tube (3EO Key) where reverse transcription, Loop-Mediated Isothermal DNA Amplifications (LAMP) processing and sequence-specific probe technologies to detect segments of the SARS-CoV-2 genome are managed automatically by the 3EO Health Cube test reader.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals suspected of COVID-19 disease by a healthcare provider or individuals who have tested positive within the past 7 calendar days with a confirmed positive COVID-19 test
2. Individuals able to self-administer the investigational test either upon themselves or upon their child (under sixteen (16) years of age) as a parent or guardian
3. Individuals willing and able to provide informed consent or obtain consent from legal authorized representative (LAR)

Exclusion Criteria:

1. If symptomatic, individuals with self-declared symptoms greater than 7 days (plus/minus 1 day, if symptoms start not definite)
2. Unable to provide consent or obtain consent from a LAR
3. Unwilling or unable to collect all sample types
4. Enrolled in a study to evaluate an investigational drug
5. Eating/drinking/smoking 30 minutes prior to specimen collection
6. Prisoner or under incarceration
7. Have contraindications to the collection of nasal specimens from the nares/nostrils, such as but not limited to nasal ulcers or nasal surgery within 3 months prior to sample collection

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Correlation of the 3EO Health SARS-CoV-2 standard of care (PCR) Zymo rRT-PCR results of the anterior nare sample. | 1-16 weeks
  The primary endpoints of this study will be the correlation of the 3EO Health SARS-CoV-2 OTC At Home Test results from nasal samples to the comparator, standard of care (PCR) Zymo rRT-PCR results of the anterior nare sample.

CONTACTS AND LOCATIONS:
Overall Officials: Jerika Acosta, Study Director — Medicept Inc.
Locations (5):
- United States (5):
  - Sarkis Clinical Trials, Gainesville, Florida
  - I.V.A.M. Clinical & Investigational Center, Miami, Florida
  - Sunrise Research Institute, Sunrise, Florida
  - Vytalus Medical Atascocita, Humble, Texas
  - Vytalus Medical, Kingwood, Texas

IPD SHARING:
Plan to Share IPD: No